CLINICAL TRIAL: NCT03814421
Title: Effect of Intermittent Versus Continuous Intravenous Pantoprazole for Prevention of Bleeding After Endoscopic Therapy of Bleeding Peptic Ulcers
Brief Title: Efficacy of Low Dose Intravenous Proton Pump Inhibitor for Peptic Ulcer Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Changwon Hospital (Other)
Responsible Party: Principal Investigator, Jung Won Lee, Professor, Samsung Changwon Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-SCMC-008-00
Record Dates: First submitted 2019-01-07; First posted 2019-01-24 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Peptic Ulcer Hemorrhage; Peptic Ulcer, Acute With Hemorrhage; Peptic Ulcer; Proton Pump Inhibitor Overdose
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Peptic Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose intermittent (Experimental): Pantoprazole 40mg as a bolus injection daily for 72hours
  Interventions: Drug: intermittent (40mg as a bolus injection daily for 72hours)
- High dose continous (Active Comparator): Pantoprazole 40mg as a bolus injection followed by continuous infusion at 8mg/hr for 72hours
  Interventions: Drug: intermittent (40mg as a bolus injection daily for 72hours)

INTERVENTIONS:
Drug: intermittent (40mg as a bolus injection daily for 72hours) — Current guidelines recommend an intravenous bolus dose of a proton pump inhibitor(PPI) followed by continuous PPI infusion after endoscopic therapy in patients with high-risk bleeding peptic ulcers. However, recent many studies suggests intermittent low dose PPI infusion might have equal efficacy at preventing peptic ulcer hemorrhage recurrence. So, the present investigator assumed that intermittent administration of proton pump inhibitor will not be different from administration of continuous proton pump inhibitor for the prevention of rebleeding in patients with peptic ulcer bleeding. Also, intermittent proton pump inhibitor administration in patients with high risk of rebleeding (Rockall score 6 points or more) will not be different from prevention of rebleeding compared with continuous proton pump inhibitor administration.

SUMMARY:
We prepare this study to compare the efficacy of intermittent intravenous PPI infusion (relatively low dose PPI therapy) than continous PPI infusion method. Our hypothesis is that intermittent (40mg as a bolus injection daily for 72 hours) PPI therapy is not inferior to conventional high dose therapy.

DETAILED DESCRIPTION:
Background Current guidelines recommend an intravenous bolus dose of a proton pump inhibitor(PPI) followed by continuous PPI infusion after endoscopic therapy in patients with high-risk peptic ulcer bleeding. However, intermittent PPI have not been inferior to continuous PPI infusion regimens in recent studies.

Objective The aim of this study was to compare the effect of intermittent (40mg as a bolus injection daily for 72hours) versus continuous (40mg as a bolus injection followed by continuous infusion at 8mg/hr for 72hours) intravenous pantoprazole for prevention of bleeding after endoscopic therapy of peptic ulcer bleeding. Also, the same comparison was performed in high-risk patients (Rockall scores ≥6).

Methods This single center cross-sectional study was conducted from january 2010 through december 2013. Patients who presented with overt or suspected upper gastrointestinal bleeding based on hematemesis and/or melena were eligible. These eligible patients were required to have a peptic ulcer with bleeding on emergency endoscopy performed within 24 hours after hospitalization. Exclusion criteria were refusal of endoscopy, gastrointestinal malignancy, Mallory-Weiss syndrome, variceal bleeding, bleeding d/t endoscopic procedure, small bowel bleeding, serious medical disease, etc. Demographic and medical data were obtained from the patients' medical records. Current or past history of medical diagnosis and drug history were also recorded. Statistical analysis performed using SPSS 21.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who had undergone gastroscopy for melena, hematochezia or hematemesis due to bleeding peptic ulcers were eligible. These eligible patients were required to have a peptic ulcer with bleeding on emergency endoscopy performed within 24 hours after hospitalization

Exclusion Criteria:

* refusal of endoscopy, gastrointestinal malignancy, Mallory-Weiss syndrome, variceal bleeding, bleeding d/t endoscopic procedure, small bowel bleeding, serious medical disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
rebleeding rates within 7 days | Within 7 days from enrollment of patient
  Rebleeding was defined that endoscopy confirms that the bleeding is completely controlled and the following outcomes occur after initial vital signs are stabilized.
  1. when a new hematemesis, hematochezia, occurs.
  2. melena occurs and blood pressure decreases (less than 90 mmHg) or pulse rate increase (110 beats per minute) or hemoglobin decline (greater than 3 g / dL) within 24 hours.

SECONDARY OUTCOMES:
Transfusion requirement | within 7 days from enrollment of patient
  The amount of transfusion that occurred during the period when the patient was in hospital was recorded as unit.
Hospital stay | within 1 years from enrollment of patient
  length of hospital stay - From the day the patient visits the emergency room to the day when the patient gets discharged
Death related with Upper GI bleeding | within 1 years from enrollment of patient
  All-cause or bleeding-related mortality was observed within 1 year of patient enrollment.
Operation d/t Upper GI bleeding | within 1 years from enrollment of patient
  This result is defined as exploratory laparatomy associated with peptic ulcer bleeding, gastric and duodenal resection anastomosis, and vagotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Changwon Hospital, Changwon, Gyeongsangnam-do, South Korea

REFERENCES:
- [Background] Sung JJ, Chiu PW, Chan FKL, Lau JY, Goh KL, Ho LH, Jung HY, Sollano JD, Gotoda T, Reddy N, Singh R, Sugano K, Wu KC, Wu CY, Bjorkman DJ, Jensen DM, Kuipers EJ, Lanas A. Asia-Pacific working group consensus on non-variceal upper gastrointestinal bleeding: an update 2018. Gut. 2018 Oct;67(10):1757-1768. doi: 10.1136/gutjnl-2018-316276. Epub 2018 Apr 24. PMID 29691276
- [Result] Sreedharan A, Martin J, Leontiadis GI, Dorward S, Howden CW, Forman D, Moayyedi P. Proton pump inhibitor treatment initiated prior to endoscopic diagnosis in upper gastrointestinal bleeding. Cochrane Database Syst Rev. 2010 Jul 7;2010(7):CD005415. doi: 10.1002/14651858.CD005415.pub3. PMID 20614440
- [Result] Cook D, Guyatt G. Prophylaxis against Upper Gastrointestinal Bleeding in Hospitalized Patients. N Engl J Med. 2018 Jun 28;378(26):2506-2516. doi: 10.1056/NEJMra1605507. No abstract available. PMID 29949497